CLINICAL TRIAL: NCT02042196
Title: Biological Mechanisms of Vascular Dysfunction With Age and Estrogen Deficiency
Brief Title: Sex Hormones and Atherosclerosis Prevention in Perimenopausal Women
Acronym: SHAPE2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 06-0537 SHAPE2; R56HL114073-06A1 (NIH)
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Menopause; Aging
Keywords: endothelial function; women; estrogen deficiency; sex hormones; adiposity; oxidative stress; antioxidants
MeSH Terms: conditions — Obesity | interventions — sapropterin; cetrorelix; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre or Early perimenopausal 1 (Experimental): Baseline experiment: Subjects randomized to either 1) KUVAN (10mg/kg body weight) crossover to placebo OR 2) placebo crossover to KUVAN
  Hormone modification: GnRH antagonist with Cetrotide (0.25mg/d) + placebo transdermal patch, then subjects randomized again to either 1) KUVAN crossover to placebo OR 2) placebo crossover to KUVAN
  Interventions: Drug: KUVAN; Drug: Placebo; Drug: Cetrotide; Drug: Placebo transdermal patch
- Pre or Early Perimenopausal 2 (Experimental): Baseline experiment: Subjects randomized to either 1) KUVAN crossover to placebo OR 2) placebo crossover to KUVAN
  Hormone modification: Estrogen add-back with Cetrotide + Climara (0.075mg/d), then subjects randomized again to either 1) KUVAN crossover to placebo OR 2) placebo crossover to KUVAN
  Interventions: Drug: KUVAN; Drug: Placebo; Drug: Cetrotide; Drug: Climara
- Late Perimenopausal and Postmenopausal (Experimental): Subjects randomized to either 1) KUVAN crossover to placebo OR 2) placebo crossover to KUVAN
  No hormone modification.
  Interventions: Drug: KUVAN; Drug: Placebo

INTERVENTIONS:
Drug: KUVAN — KUVAN will be given orally at 10mg/kg dose per body weight. KUVAN will be dissolved in 4-8oz water and consumed within 15 minutes.
  Other Names: Tetrahydrobiopterin or BH4
Drug: Placebo — Placebo pills designed to match the dissolvable KUVAN pills
  Other Names: Control
Drug: Cetrotide — Cetrotide (0.25mg/d) will be taken daily for 10 days via abdominal subcutaneous injection.
  Other Names: Cetrorelix acetate
  Arms: Pre or Early Perimenopausal 2; Pre or Early perimenopausal 1
Drug: Climara — 0.075mg/d transdermal patch will be placed on skin.
  Other Names: Estradiol transdermal patch
  Arms: Pre or Early Perimenopausal 2
Drug: Placebo transdermal patch — Inactive transdermal patch
  Other Names: Control
  Arms: Pre or Early perimenopausal 1

SUMMARY:
As women get older and go through menopause, levels of the female reproductive hormone estradiol decrease to low levels. Also with aging, the functioning of the arteries declines. Over time this vascular dysfunction can lead to health problems such as high blood pressure and heart disease. This study is being done to help determine what causes arteries to become unhealthy in postmenopausal women, who have low levels of the female reproductive hormone estradiol. In this study we will test whether low levels of tetrahydrobiopterin (BH4), a natural substance in the body that can cause the arteries to expand, explains why arteries become unhealthy in women with low levels of estradiol. To answer this question, we will study how vascular function changes with a medication that causes a short-term increase in BH4 levels when estradiol is lowered with a medication, compared to when estradiol is normal. We will also determine whether the administration of the antioxidant vitamin C, along with the medication to increase BH4 levels, will normalize vascular health in perimenopausal and postmenopausal women, and in women who have their estradiol levels lowered.

DETAILED DESCRIPTION:
Endothelial dysfunction, featuring reduced vascular endothelial-dependent dilation (EDD), is a significant predictor of cardiovascular (CV) events. Reduced EDD is characterized by the loss of nitric oxide (NO) production. EDD declines with aging in women at a slower rate compared to men but rapidly declines after menopause and quickly catches up to men, suggesting a beneficial effect of estrogen (E2). Our research has investigated the mechanisms underlying endothelial protection of E2 including how hormonal fluctuations during the peri-to early postmenopausal years contribute to endothelial dysfunction, and how these hormonal changes might interact with aging. Using a well described experimental model (systemic infusion of ascorbic acid; AA) to acutely reduce reactive oxygen species (ROS), our preliminary findings implicate oxidative stress as an underlying mechanism explaining the impaired EDD during the menopausal transition. Specifically we found improved EDD in response to AA in late peri- and postmenopausal women but not in pre- or early perimenopausal women. These data indicate that E2 may protect the vasculature from free radical injury during pre- and early perimenopausal years. In support of this concept, we demonstrated that AA can reverse the decrease in EDD that occurs in the setting of short-term E2 deficiency (3-days of gonadotropin releasing hormone antagonist; GnRHant) in pre-and early perimenopausal women.

Tetrahydrobiopterin (BH4) is a critical co-factor in the production of NO by endothelial nitric oxide synthase (eNOS), and in the face of deficient levels, uncoupling of eNOS results in the production of ROS instead of NO. Whether the increased ROS and impaired EDD that occurs during the peri- and early postmenopausal periods is associated with reduced vascular BH4 is at present unknown. However, our finding that AA could not improve the reduced EDD found in early perimenopausal women or restore EDD in peri-and postmenopausal women to premenopausal levels, indicates that other sources of ROS or causes of low NO are involved in the impaired EDD across the stages of the menopause transition and aging in women. In vitro studies demonstrate that the co-administration of BH4 and AA completely prevents the eNOS uncoupling and decreased NO production in endothelial cells treated with a peroxynitrite (ONOO-) donor, compared to administering either one alone. The global aim of this renewal is to follow-up on our previous findings and to determine the role of BH4 as a mediator of endothelial dysfunction [across the stages of the menopausal transition and aging in women. This global aim will be addressed by 3 specific aims (SA). Using a cross-sectional design, SA1 will measure EDD in healthy pre-, peri- and postmenopausal women: 1) under basal conditions; and 2) following an acute increase in BH4. SA2 will expand on the cross-sectional comparisons via short-term (10 days) ovarian suppression (GnRhant) in pre-and early perimenopausal women to isolate the age-independent effects of E2. SA3 will examine whether co-administration of BH4 and AA fully restore youthful EDD in peri-and postmenopausal women.

SA1: To determine the possible mechanistic involvement of BH4 deficiency in the decline in endothelial function during the peri-and early postmenopausal period and its potential relation to oxidative stress. This will be assessed by comparing brachial artery EDD and plasma and endothelial cell markers of oxidative stress and NO (see methods for details) in healthy pre-, peri-and postmenopausal women: 1) under basal conditions; and 2) in response to acute oral BH4 (vs PL) supplementation.

Hypothesis1 (H1): a) EDD will increase in response to BH4 in early peri, late peri and postmenopausal women but not premenopausal women. b) The increase in EDD in response to BH4 will be associated with a decrease in plasma markers of oxidative stress. c) The reduced EDD in peri- and postmenopausal women will be associated with lower endothelial cell markers of NO and higher oxidative Stress.

SA2: To determine whether the decrease in EDD in response to acute ovarian suppression in pre- and early perimenopausal women is related to reduced BH4 bioavailability and elevated markers of oxidative stress. This will be assessed by comparing EDD and plasma markers of oxidative stress after acute oral supplementation of BH4 (or PL) following either acute ovarian suppression with (GnRHant+E2) or without (GnRHant+PL) E2 add-back. Additionally, endothelial cell protein expression of markers of BH4 biosynthesis and oxidative stress will be measured before and after the suppression/add-back paradigm.

H2: a) The expected decrease in EDD and increase in plasma oxidative stress markers following acute ovarian suppression will be mitigated in the groups treated with oral BH4 (GnRHant+PL+BH4); there will be little or no effect of the addition of BH4 to the E2 add-back group. b) Ovarian suppression alone will reduce endothelial protein markers of BH4 biosynthesis and will increase markers of oxidative stress. These changes will not be observed following ovarian suppression with E2 add-back and oral BH4. These sets of experiments will provide evidence that the oxidative stress-related decrease in EDD in response to E2 suppression is in part, related to decreased BH4 bioavailability.

SA3: To determine whether the co-administration of BH4 with AA will completely restore EDD in peri-and postmenopausal women, and in early perimenopausal women following ovarian suppression.

H3: The co-administration of BH4 with AA will restore EDD to premenopausal levels a) in peri-and postmenopausal women, and b) in early perimenopausal following acute ovarian suppression.

ELIGIBILITY:
Inclusion Criteria:

* age criteria established for pre-, peri- and postmenopausal women, and if postmenopausal at least 1 year beyond menopause
* resting blood pressure <140/90 mmHg 81; 2) plasma glucose concentrations <110 mg/dl under fasting conditions
* sedentary or recreationally active (<3 days of vigorous aerobic exercise)
* no use of OCs, HT, or other medications that might influence cardiovascular function
* nonsmokers
* no use of vitamin supplements, NSAIDS or willing to stop use for duration of the study
* not taking any other medications that would interact with cetrotide, E2 patch, or Kuvan® to confound interpretation of results

Exclusion Criteria:

* history of or active estrogen-dependent neoplasms, acute liver or gallbladder disease, vaginal bleeding, venous thromboembolism, hypertriglyceridemia, and CVD
* known allergy to transdermal patch, GnRHant (i.e., hypersensitivity to cetrorelix, extrinsic peptide hormones, mannitol, GnRH, benzyl alcohol - the vehicle for injection of cetrorelix), or KUVAN
* history of stomach ulcer or bleeding
* other contraindications to HRT, GnRHant, and KUVAN (i.e., taking Levodopa, medications that can inhibit folate metabolism including methotrexate)
* pregnant or currently breastfeeding
* Other conditions for which individuals will be excluded from the study include: diabetes, active infection, history of seizures or disease that affects the nervous system, sepsis or an abnormal resting ECG

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery flow-mediated dilation | 4-5 years

SECONDARY OUTCOMES:
Change in carotid artery compliance and endothelial cell protein expression | 4-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Moreau, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States